CLINICAL TRIAL: NCT03038464
Title: Benefit of Synovial Aspiration and Serological Testing in Two-stage Revision Arthroplasty of Prosthetic Joint Infection
Brief Title: Synovial Aspiration and Serological Testing in Two-stage Revision Arthroplasty of Prosthetic Joint Infection
Acronym: SyPJI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Harrasser, Principal Investigator, Technical University of Munich
Other Study IDs: 445/21
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-01

CONDITIONS: Diagnosis Prosthetic Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Synovial biopsy — Biopsy of jint prior reimplantation of new joint prosthesis

SUMMARY:
The two-stage protocol is gold standard in terms of infection control treating prosthetic joint infections of total hip and total knee arthroplasty. The antibiotic pause for diagnostic reasons before reconstruction (stage two) is discussed concerning persistence of infection and development of resistant bacterial strains. Serological markers and synovial analysis are common use to exclude persistence of infection.

The investigators therefore asked 1) is the serological testing of c-reactive protein and leukocytes a valuable tool to predict a persistence of infection and 2) what is the role of synovial aspiration of PMMA Spacers on hip and knee joints.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periprostheitc joint infection

Exclusion Criteria:

* Reinfection in history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with periprostheitc joint infection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Reinfection rate | 2 years
  Reinfection rate after reimplantation of joint prosthesis

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided